CLINICAL TRIAL: NCT02623140
Title: Randomized Comparison of a Polymer-Free Biolimus-eluting BIOFREEDOM Stent With a Biodegradable-Polymer Sirolimus-eluting ORSIRO Stent in Patients Treated With Percutaneous Coronary Intervention
Brief Title: BIOFREEDOM Stent Versus ORSIRO Stent: SORT OUT IX
Acronym: SORT OUT IX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lisette Okkels Jensen, MD DMSci PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SORT OUT IX
Record Dates: First submitted 2015-11-30; First posted 2015-12-07 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Ischaemic Heart Disease
Keywords: Coronary drug eluting stents; Outcomes
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biofreedom (Experimental): Biofreedom stent treatment at index procedure
  Interventions: Device: Biofreedom
- Orsiro (Active Comparator): Orsiro stent treatment at index procedure
  Interventions: Device: Orsiro

INTERVENTIONS:
Device: Biofreedom — PCI with Biofreedom stent
  Arms: Biofreedom
Device: Orsiro — PCI with Orsiro stent
  Arms: Orsiro

SUMMARY:
The aim of the Danish Organization for Randomized Trials with Clinical Outcome (SORT OUT) is to compare the safety and efficacy of the polymer-free Biolimus-eluting BIOFREEDOM stent with a biodegradable-polymer Sirolimus-eluting ORSIRO stent in a population-based setting, using registry detection of clinically driven events

DETAILED DESCRIPTION:
SORT OUT IX is a randomized, multicenter, all-comer, two-arm, non-inferiority trial comparing the polymer-free Biolimus-eluting BIOFREEDOM stent with a biodegradable-polymer Sirolimus-eluting ORSIRO stent in treating atherosclerotic coronary artery lesions.

Patients will be enrolled by the investigators and randomly allocated to treatment groups after diagnostic coronary angiography and before percutaneous coronary intervention. Block randomization by centre (permuted blocks of random sizes (2/4/6)) will be used to assign patients in a 1:1 ratio to receive the polymer-free Biolimus-eluting BIOFREEDOM stent (Biosensors) or the biodegradable-polymer Sirolimus-eluting ORSIRO stent (Biotronik). A web based Trial Partner randomization system will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over with chronic stable coronary artery disease or acute coronary syndromes, and at least one coronary artery lesion with more than 50% diameter stenosis, requiring treatment with a drug-eluting stent.

Exclusion Criteria:

* Life expectancy of less than one year; an allergy to aspirin, clopidogrel, ticagrelor, prasugral, biolimus or sirolimus; participation in another randomized trial; or inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3150 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure | 12 months
  Primary endpoint assessed after 12 months

SECONDARY OUTCOMES:
Target lesion failure | 2 year, 3 year, 4 year, 5 year
  Target lesion failure will be assessed yearly up to 5 years after index procedure
Stent thrombosis | 1 year, 2 years, 3 years, 4 years, 5 years
  Stent thrombosis will be assessed yearly up to 5 years after index procedure
Myocardial infarction | 1 year, 2 years, 3 years, 4 years, 5 years
  Myocardial infarction will be assessed yearly up to 5 years after index procedure
Cardiac death | 1 year, 2 years, 3 years, 4 years, 5 years
  Cardiac death will be assessed yearly up to 5 years after index procedure
All cause mortality | 1 year, 2 years, 3 years, 4 years, 5 years
  All cause mortality will be assessed yearly up to 5 years after index procedure
Target lesion revascularization | 1 year, 2 years, 3 years, 4 years, 5 years
  Target lesion revascularization will be assessed yearly up to 5 years after index procedure
Target vessel revascularization | 1 year, 2 years, 3 years, 4 years, 5 years
  Target vessel revascularization will be assessed yearly up to 5 years after

CONTACTS AND LOCATIONS:
Overall Officials: Lisette Okkels Jensen, MD DMSci PhD, Study Chair — Odense University Hospital; Evald H Christiansen, MD PhD, Study Chair — Aarhus University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Jensen Lisette Okkels, Maeng M, Raungaard B, Kahlert J, Ellert J, Jakobsen L, Villadsen AB, Veien KT, Kristensen SD, Ahlehoff O, Carstensen S, Christensen MK, Terkelsen CJ, Engstroem T, Hansen KN, Botker HE, Aaroe J, Thim T, Thuesen L, Freeman P, Aziz A, Eftekhari A, Junker A, Jensen SE, Lassen JF, Hansen HS, Christiansen EH; Sort Out IX Study Group. Randomized Comparison of the Polymer-Free Biolimus-Coated BioFreedom Stent With the Ultrathin Strut Biodegradable Polymer Sirolimus-Eluting Orsiro Stent in an All-Comers Population Treated With Percutaneous Coronary Intervention: The SORT OUT IX Trial. Circulation. 2020 Jun 23;141(25):2052-2063. doi: 10.1161/CIRCULATIONAHA.119.040241. Epub 2020 May 21. PMID 32434381
- [Derived] Jensen LO, Maeng M, Raungaard B, Engstrom T, Hansen HS, Jensen SE, Botker HE, Kahlert J, Lassen JF, Christiansen EH. Comparison of the polymer-free biolimus-coated BioFreedom stent with the thin-strut biodegradable polymer sirolimus-eluting Orsiro stent in an all-comers population treated with percutaneous coronary intervention: Rationale and design of the randomized SORT OUT IX trial. Am Heart J. 2019 Jul;213:1-7. doi: 10.1016/j.ahj.2019.02.017. Epub 2019 Mar 14. PMID 31055192